CLINICAL TRIAL: NCT03578562
Title: A Prospective Cohort Study on Targeted Exercise and Changes in Femoroacetabular Impingement in Symptomatic Patients With Acetabular Retroversion (TILT-FAI)
Brief Title: Targeted Exercise and Changes in Femoroacetabular Impingement in Symptomatic Patients With Acetabular Retroversion
Acronym: TILT-FAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); University College Absalon. Region of Zealand, Denmark (Unknown); The Danish Rheumatism Association (Other); Vanfoerefonden, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1- Brekke
Record Dates: First submitted 2018-05-09; First posted 2018-07-06 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Acetabular Dysplasia
Keywords: Femoroacetabular Impingement; Anterior Pelvic Tilt
MeSH Terms: conditions — Hip Dislocation; Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted training intervention (Experimental): An 8-week progressive homebased training intervention with supervised booster-sessions
  Interventions: Other: Targeted training intervention

INTERVENTIONS:
Other: Targeted training intervention — An 8-week progressive homebased training intervention with supervised booster-sessions

SUMMARY:
The objective of this study is to investigate the effectiveness of an 8-week home-based targeted training intervention aiming at reducing FAI related pain, anterior pelvic tilt and improve hip joint function in a cohort of 40 patients (18 to 40 years), with acetabular retroversion and anterior pelvic tilt not eligible for surgery (Ganz osteotomy) from the hospital outpatient clinic.

DETAILED DESCRIPTION:
Acetabular retroversion is a variation of hip dysplasia, reported in the normal population from 6 % to 48 %, enhancing the risk of femoroacetabular impingement (FAI) in especially hip flexion and is associated with pain, reduced level of function, decreased health-related quality of life and early development of osteoarthritis (OA) of the hip. A higher degree of anterior pelvic tilt increases the risk of FAI and especially in standing, sitting and squatting positions it has been found to correlate with FAI. Periacetabular osteotomy (Ganz osteotomy) is performed as a surgical joint preserving reorientation of the entire acetabulum with a subsequently long period of rehabilitation. There is currently no existing alternative (i.e. non-surgical) treatment to surgery for this patient group. Therefore, the objective of this study is to test a targeted training intervention aiming at reducing anterior pelvic tilt and improve hip joint function in patients with symptomatic acetabular retroversion.

A prospective cohort study of 40 patients will undergo an 8-week targeted exercise intervention executed as progressive home-based training with supervised booster-sessions. Patients (18 to 40 years) with acetabular retroversion and anterior pelvic tilt not eligible for surgery (Ganz osteotomy) will be recruited from the outpatient clinic.

Time points for testing are at 1) minus 8-weeks (beginning of control-period) 2) baseline (beginning of training period) 3) plus 8-weeks (end of training period) and 4) plus 26 weeks from baseline (follow up).

The primary outcome measure is self-perceived level of hip related pain (HAGOS questionnaire subscale). Secondary outcome measures are self-perceived level of function and quality of life (remaining HAGOS-subscales), EQ-5D-3Levels questionnaire and radiographic degree of pelvic tilt in standing posture (EOS-scanning). Explorative outcome measures include additional radiographic measurements, patient-reported outcome measurements (PROM´s), functional testing and physical performance. The primary endpoint for assessing the outcome of the intervention will be 8 weeks after start of intervention. At 26-week follow up, only the PROM´s will be applied. All participants must fill in a mandatory exercise related dairy concerning adherence, level of pain and potential adverse events.

The study is approved by the Regional Committees on Health Research Ethics for Southern Denmark, Project ID: S-20160072 Forty participants in total will be enrolled from the hip outpatient clinic at Odense University Hospital, Denmark. Paired means sample size calculation = 36 (10 % pre-posttest difference on HAGOS pain-subscale, SD=20.6, alpha = 0.05, power = 80 %), plus 10 % dropout = 4.

A list generated of 20 randomly found numbers from 1-40 will be used to select participants to be investigated in the motion laboratory. The number on the list corresponds to the order the participants are recruited into the study. In the motion laboratory, the explorative outcomes Functional testing (3D motion capture) and Physical performance (isometric muscle strength, joint range-of-motion, and single-leg hop for distance) will be tested.

To our knowledge, this is the first study investigating a targeted training intervention aiming at reducing FAI related pain, anterior pelvic tilt and improve hip joint function in patients with acetabular retroversion. Consequently, the study will provide knowledge that may help to develop non-surgical treatment strategies for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed from a standard standing anterior-posterior pelvic radiograph with acetabular retroversion due to cross-over-sign and posterior-wall-sign
* Not eligible for Ganz osteotomy
* Ability to take part in the intervention

Exclusion Criteria:

* Having a Pelvic Tilt Ratio greater than 0.5, (the height of the obturator foramen divided by the height of the lesser pelvis) indicating posterior pelvic tilt, assessed from a standard standing AP-pelvic radiograph
* Radiographic sign of hip osteoarthritis (< 2mm. joint space),
* Previous lumbar, pelvic or hip related operations
* Conditions not allowing exercise therapy
* Body mass index (BMI) above 35
* Not understanding spoken and/or written Danish language

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
HAGOS questionnaire (pain subscale) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention) and 26 weeks (follow up from baseline)
  Change in The Copenhagen Hip and Groin Outcome Score (HAGOS) questionnaire pain subscale.
  Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4, where 0 indicates no problem. The scores from each subscale are calculated as the sum of the items included. Raw scores are then transformed to a 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.

SECONDARY OUTCOMES:
HAGOS questionnaire (the remaining five subscales) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention) and 26 weeks (follow up from baseline)
  Change in the remaining five HAGOS-subscales (Symptoms, Physical function in daily living, Physical function in Sport and Recreation, Participation in Physical Activities and hip and/or groin-related Quality of Life).
  Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4, where 0 indicates no problem. The scores from each subscale are calculated as the sum of the items included. Raw scores are then transformed to a 0-100 scale, with zero representing extreme hip and/or groin problems and 100 representing no hip and/or groin problems.
EQ-5D-3Levels questionnaire | Minus 8-weeks (control), baseline, 8-weeks (post-intervention) and 26 weeks (follow up from baseline).
  Change in the European Quality of Life - 5 Dimensions (EQ-5D-3Levels) questionnaire, Danish version. For each dimension (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression) standardized answer options are divided in levels of perceived problems (3 Likert boxes): Level 1: indicating no problem, Level 2: indicating some problems, Level 3: indicating extreme problems. A unique health state is defined by combining the selected level from each of the 5 dimensions. In addition, the overall health state the actual day is marked on a numeric scale on which the best state is marked 100 and the worst state is marked 0.
Radiographic measurement of pelvic tilt (SCJ - Symphysis distance) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in the degree of pelvic tilt measured in the frontal plane as the distance (in mm) from the sacro-coccygeal joint (SCJ) to the upper border of the pubic symphysis (standing EOS scanning)

OTHER OUTCOMES:
Global Perceived Effect anchor-question | 8-weeks (post-intervention) and 26 weeks (follow up from baseline)
  Changed from baseline on a 7-point Likert scale: ´much better, better, little better, unchanged, little worse, worse, much worse'.
Oxford 12-item Hip Score (OHS) questionnaire, Danish version | Minus 8-weeks (control), baseline, 8-weeks (post-intervention) and 26 weeks (follow up from baseline)
  Change in Oxford Hip Score (OHS) questionnaire. Standardized answer options are given (5 Likert boxes) and each question gets a score from 1 to 5, where 1 indicates no problem. The score is calculated as the sum of the 12 questions. The score can therefore be 12-60. The higher the score, the lower the function level.
UCLA activity scale | Minus 8-weeks (control), baseline, 8-weeks (post-intervention) and 26 weeks (follow up from baseline).
  Change in the University of California Los Angeles activity-level rating (UCLA activity scale), Danish version. On a 10-point scale, the option is marked that matches the level of intensity and frequency of physical activity best, where 1 ="Wholly inactive: depend on others, cannot leave residence, and 10 =" Regularly participates in impact sports".
Radiographic measurement of pelvic tilt (pelvic tilt ratio) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in pelvic tilt ratio measured in the frontal plane (standing EOS scanning) and calculated as the centrally height (in mm) of the obturator foramens divided by the centrally height (in mm) of the lesser pelvis (the distance from the two lower margins of the sacroiliac joint to the upper border of the two obturator foramens).
Radiographic measurement of pelvic tilt (sagittal plane) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in pelvic tilt (in degrees) measured in the sagittal plane (standing EOS scanning) as the angle between a horizontal line and a line connecting the upper border of the symphysis with the sacral promontory.
Radiographic measurements of pelvic parameters (Pelvic Incidence) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Pelvic Incidence (in degrees) measured as the angle between the line joining the hip axis and the center of the S1 end-plate and the line orthogonal to the S1 end-plate (standing EOS scanning)
Radiographic measurements of pelvic parameters (Pelvic Tilt) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Pelvic Tilt (in degrees) measured as the angle between the line joining the hip axis and the center of the S1 end-plate and a reference vertical line (standing EOS scanning)
Radiographic measurements of pelvic parameters (Sacral Slope) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Sacral Slope (in degrees) measured as the angle between the line along the S1 end-plate and a reference horizontal line (standing EOS scanning)
Radiographic parameters of acetabular retroversion (Cross-Over Sign) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Cross-Over Sign (yes/no) (standing EOS scanning)
Radiographic parameters of acetabular retroversion (Cross-Over Ratio) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Acetabular Cross-Over Ratio (percent) (standing EOS scanning)
Radiographic parameters of acetabular retroversion (Posterior Wall Sign) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Posterior Wall Sign (yes/no) (standing EOS scanning)
Radiographic parameters of acetabular retroversion (Posterior Wall Ratio) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Posterior Wall Ratio (percent) (standing EOS scanning)
Radiographic parameters of acetabular retroversion (Ischial Spine Sign) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in Ischial Spine Sign (yes/no) (standing EOS scanning)
Physical performance (hip muscle strength) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in maximal isometric hip extension, flexion and abduction muscle strength (in Nm using dynamometry)
Physical performance (abdominal muscle strength) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in maximal isometric abdominal muscle strength (in Nm using dynamometry)
Physical performance (hip ROM) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip extension range-of-motion (in degrees using goniometry)
Physical performance (lumbar spine ROM) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in lumbar spine flexion range-of-motion (in cm. using Schobers test)
Physical performance (Single-leg hop for distance) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention).
  Change in the horizontal single-leg hop distance (in cm) from the toe in the starting position to the heel in the landing position.
Functional test (3D Gait analysis - kinetics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in peak- and mean hip joint moments (in Nm) using 3D Vicon motion capture analysis
Functional test (3D Gait analysis - kinematics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip joint range-of-motion (in degrees) using 3D Vicon motion capture analysis
Functional test (3D deep squat analysis - kinetics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in peak- and mean hip joint moments (in Nm) using 3D Vicon motion capture analysis
Functional test (3D deep squat analysis - kinematics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip joint range-of-motion (in degrees) using 3D Vicon motion capture analysis
Functional test (3D deep squat analysis, with heel support - kinetics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in peak- and mean hip joint moments (in Nm) using 3D Vicon motion capture analysis
Functional test (3D deep squat analysis, with heel support - kinematics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip joint range-of-motion (in degrees) using 3D Vicon motion capture analysis
Functional test (3D counter movement jump analysis, unilateral - kinetics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in peak- and mean hip joint moments (in Nm) using 3D Vicon motion capture analysis
Functional test (3D counter movement jump analysis, unilateral - kinematics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip joint range-of-motion (in degrees) using 3D Vicon motion capture analysis
Functional test (3D counter movement jump analysis, bilateral - kinetics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in peak- and mean hip joint moments (in Nm) using 3D Vicon motion capture analysis
Functional test (3D counter movement jump analysis, bilateral - kinematics) | Minus 8-weeks (control), baseline, 8-weeks (post-intervention)
  Change in hip joint range-of-motion (in degrees) using 3D Vicon motion capture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anders F Brekke, PT, MSc, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark - Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized and stored in a encrypted Sharepoint folder. With permission from the scientific person responsible for the present study, the data will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion February 2020 all data will be anonymized and stored in a secure Sharepoint folder indefinitely.
Access Criteria: The Sharepoint folder is hosted by Odense University Hospital, Region Southern Denmark. Only employees from the Orthopaedic Research unit at Odense University Hospital can access the folder using individual log in codes.

REFERENCES:
- [Background] Reynolds D, Lucas J, Klaue K. Retroversion of the acetabulum. A cause of hip pain. J Bone Joint Surg Br. 1999 Mar;81(2):281-8. doi: 10.1302/0301-620x.81b2.8291. PMID 10204935
- [Background] Ezoe M, Naito M, Inoue T. The prevalence of acetabular retroversion among various disorders of the hip. J Bone Joint Surg Am. 2006 Feb;88(2):372-9. doi: 10.2106/JBJS.D.02385. PMID 16452750
- [Background] Werner CM, Copeland CE, Ruckstuhl T, Stromberg J, Seifert B, Turen CH. Prevalence of acetabular dome retroversion in a mixed race adult trauma patient population. Acta Orthop Belg. 2008 Dec;74(6):766-72. PMID 19205323
- [Background] Langlais F, Lambotte JC, Lannou R, Gedouin JE, Belot N, Thomazeau H, Frieh JM, Gouin F, Hulet C, Marin F, Migaud H, Sadri H, Vielpeau C, Richter D. Hip pain from impingement and dysplasia in patients aged 20-50 years. Workup and role for reconstruction. Joint Bone Spine. 2006 Dec;73(6):614-23. doi: 10.1016/j.jbspin.2006.09.001. Epub 2006 Oct 25. PMID 17137820
- [Background] Rylander JH, Shu B, Andriacchi TP, Safran MR. Preoperative and postoperative sagittal plane hip kinematics in patients with femoroacetabular impingement during level walking. Am J Sports Med. 2011 Jul;39 Suppl:36S-42S. doi: 10.1177/0363546511413993. PMID 21709030
- [Background] Clohisy JC, Baca G, Beaule PE, Kim YJ, Larson CM, Millis MB, Podeszwa DA, Schoenecker PL, Sierra RJ, Sink EL, Sucato DJ, Trousdale RT, Zaltz I; ANCHOR Study Group. Descriptive epidemiology of femoroacetabular impingement: a North American cohort of patients undergoing surgery. Am J Sports Med. 2013 Jun;41(6):1348-56. doi: 10.1177/0363546513488861. Epub 2013 May 13. PMID 23669751
- [Background] Ganz R, Parvizi J, Beck M, Leunig M, Notzli H, Siebenrock KA. Femoroacetabular impingement: a cause for osteoarthritis of the hip. Clin Orthop Relat Res. 2003 Dec;(417):112-20. doi: 10.1097/01.blo.0000096804.78689.c2. PMID 14646708
- [Background] Ross JR, Nepple JJ, Philippon MJ, Kelly BT, Larson CM, Bedi A. Effect of changes in pelvic tilt on range of motion to impingement and radiographic parameters of acetabular morphologic characteristics. Am J Sports Med. 2014 Oct;42(10):2402-9. doi: 10.1177/0363546514541229. Epub 2014 Jul 24. PMID 25060073
- [Background] Riviere C, Hardijzer A, Lazennec JY, Beaule P, Muirhead-Allwood S, Cobb J. Spine-hip relations add understandings to the pathophysiology of femoro-acetabular impingement: A systematic review. Orthop Traumatol Surg Res. 2017 Jun;103(4):549-557. doi: 10.1016/j.otsr.2017.03.010. Epub 2017 Apr 1. PMID 28373141
- [Background] Ganz R, Klaue K, Vinh TS, Mast JW. A new periacetabular osteotomy for the treatment of hip dysplasias. Technique and preliminary results. Clin Orthop Relat Res. 1988 Jul;(232):26-36. PMID 3383491
- [Background] Schwarz T, Benditz A, Springorum HR, Matussek J, Heers G, Weber M, Renkawitz T, Grifka J, Craiovan B. Assessment of pelvic tilt in anteroposterior radiographs by means of tilt ratios. Arch Orthop Trauma Surg. 2018 Aug;138(8):1045-1052. doi: 10.1007/s00402-018-2931-z. Epub 2018 Apr 12. PMID 29651575

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03578562/SAP_000.pdf